CLINICAL TRIAL: NCT05795192
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Dosing, Dose-escalation, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, PK/PD, Food Effect, and Ethnicity Effect of SB17170 in Healthy Adult Subjects
Brief Title: SB17170 Phase1 Trial in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SPARK Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMARTT-002
Record Dates: First submitted 2023-02-27; First posted 2023-04-03 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Safety Issues; Tolerability; Pharmacokinetics; Pharmacodynamics
Keywords: HMGB1

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Block randomized, double-blind design controlling with IWRS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- SB17170 of 50mg, Single dose (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 50mg capsule, QD for 1 day(single).
  Interventions: Drug: SB17170
- Placebo of 50mg, Single dose (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 50mg, QD for 1 day(single).
  Interventions: Drug: Placebo
- SB17170 of 150mg, Single dose (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 100mg and 50mg capsules, QD for 1 day(single).
  Interventions: Drug: SB17170
- Placebo of 150mg, Single dose (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 100mg and 50mg capsules, QD for 1 day(single).
  Interventions: Drug: Placebo
- SB17170 of 250mg, Single dose (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg capsule, QD for 1 day(single).
  Interventions: Drug: SB17170
- Placebo of 250mg, Single dose (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 250mg capsule, QD for 1 day(single).
  Interventions: Drug: Placebo
- SB17170 of 500mg, Single dose, Food-effect (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg 2 capsules, QD for 1 day(single).
  Food-effect test for the expected efficacy dose
  * 1st period without a meal
  * Wash out period more than 7 days
  * 2nd period with a high-fat meal
  Interventions: Drug: SB17170
- Placebo of 500mg, Single dose, Food-effect (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 2 250mg 2 capsules, QD for 1 day(single).
  Food-effect test for the expected efficacy dose
  * 1st period without a meal
  * Wash out period more than 7 days
  * 2nd period with a high-fat meal
  Interventions: Drug: Placebo
- SB17170 of 1000mg, Single dose (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg 4capsules, QD for 1 day(single).
  Interventions: Drug: SB17170
- Placebo of 1000mg, Single dose (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 2 250mg 4 capsules, QD for 1 day(single).
  Interventions: Drug: Placebo
- SB17170 of 1500mg, Single dose (Experimental): Optional dose Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg 6 capsules, QD for 1 day(single).
  Interventions: Drug: SB17170
- Placebo of 1500mg, Single dose (Placebo Comparator): Optional dose Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 250mg 6 capsules, QD for 1 day(single).
  Interventions: Drug: Placebo
- SB17170 of 250mg, Multiple dose for 7days (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg, 1 capsule, QD for 7 days(multiple).
  Interventions: Drug: SB17170
- Placebo of 250mg, Multiple dose for 7days (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 250mg, 1 capsule, QD for 7 days(multiple).
  Interventions: Drug: Placebo
- SB17170 of 500mg, Multiple dose for 7days (Experimental): Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg, 2 capsules, QD for 7 days(multiple).
  Interventions: Drug: SB17170
- Placebo of 500mg, Multiple dose for 7days (Placebo Comparator): Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 250mg, 2 capsules, QD for 7 days(multiple).
  Interventions: Drug: Placebo
- SB17170 of 1000mg, Multiple dose for 7days (Experimental): Optional dose Assign 6 subjects per cohort including Korean and Caucasian. Prescribe SB17170 250mg, 4 capsules, QD for 7 days(multiple).
  Interventions: Drug: SB17170
- Placebo of 1000mg, Multiple dose for 7days (Placebo Comparator): Optional dose Assign 2 subjects per cohort including Korean and Caucasian. Prescribe Placebo 250mg, 4 capsules, QD for 7 days(multiple).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB17170 — Taking SB17170 orally once a day
  Arms: SB17170 of 1000mg, Multiple dose for 7days; SB17170 of 1000mg, Single dose; SB17170 of 1500mg, Single dose; SB17170 of 150mg, Single dose; SB17170 of 250mg, Multiple dose for 7days; SB17170 of 250mg, Single dose; SB17170 of 500mg, Multiple dose for 7days; SB17170 of 500mg, Single dose, Food-effect; SB17170 of 50mg, Single dose
Drug: Placebo — Taking Placebo orally once a day
  Arms: Placebo of 1000mg, Multiple dose for 7days; Placebo of 1000mg, Single dose; Placebo of 1500mg, Single dose; Placebo of 150mg, Single dose; Placebo of 250mg, Multiple dose for 7days; Placebo of 250mg, Single dose; Placebo of 500mg, Multiple dose for 7days; Placebo of 500mg, Single dose, Food-effect; Placebo of 50mg, Single dose

SUMMARY:
This clinical trial aims to learn about the safety, tolerability, and pharmacokinetic properties of SB17170 and its active metabolite SB1703 in single and multiple oral administration in healthy adults.

The main questions it aims to answer are the safety, tolerability, and PK characteristics of SB17170 in healthy adults.

DETAILED DESCRIPTION:
This clinical trial aims to learn about the safety, tolerability, and Pharmacokinetic properties of SB17170 and its active metabolite SB1703 in single and multiple oral administration in healthy adults.

The main questions it aims to answer are the safety, tolerability, and PK characteristics of SB17170 in healthy adults.

The second questions are

* To explore biomarkers and evaluate pharmacodynamic properties with ex-vivo test and proteome assay for SB17170
* To evaluate the effects of ethnic differences on the safety, tolerability, and pharmacokinetic properties of SB17170 in healthy Korean and Caucasian adults.
* To evaluate the effect of food between Fast and high-fat meals on safety, tolerability, and pharmacokinetic properties of SB17170 in healthy adults.

The difference between SB17170 and placebo on safety, tolerability, and PK/PD properties will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Korean or Caucasian adults between the ages of 19 and 50 as of the date of written consent
* Subjects with a body weight of 55.0 kg or more at the time of screening and a body mass index (BMI) of 18.0 kg/m2 or more and less than 30.0 kg/m2
* Written informed consent

Exclusion Criteria:

* Clinical significant medical history
* Gastrointestinal disease or past history
* Hypersensitivity or clinically significant hypersensitivity to the components of investigational drugs
* Screening test AST, ALT > ULN x 1.5 Creatinine clearance < 60mL/min/1.73m2 QTcB interval > 450 ms Serologic test positive(Hepatitis B, Hepatitis C, HIV)
* SBP <90 mmHg or >150 mmHg, DBP <60 mmHg or > 100 mmHg
* Drub abuse history
* Administration of any OTC drug, Herbal drug, Investigational medication within 2weeks
* Participation in other clinical trial within 6 months

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From Day 1 to Day 7 for Single dose, From Day 1 to Day 9 for Multiple dose
  Safety and Tolerability in healthy subjects

SECONDARY OUTCOMES:
The Area Under the Curve from dosing to the time of the last measured concentration | Baseline 0hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The area under the curve from time 0 extrapolated to infinite time(AUCinf) | Baseline 0hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The maximum (or peak) serum concentration(Cmax) | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The time to reach Cmax(Tmax) | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The Half life(t1/2) of SB17170 and active metabolite | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The ratio of oral clearance(CL/F) | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The Renal clearance(CLR) | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The volume of distribution(vd/f) | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
The ratio of unchanged drug to metabolite(Metabolic ratio) | Baseline 0 hour, 20minute, 40minute, 1hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour
  Pharmacokinetic parameter
Compare the concentrations of TNF-α between the active and placebo groups | Baseline 0 hour, 1.5hour, 24hour,
  Tumor Necrosis Factor-alpha human(TNF-α) as a Pharmacodynamic parameter
Compare the concentratiosn of Interleukin-6 between the active and placebo groups | Baseline 0 hour, 1.5hour, 24hour,
  Interleukin-6 as a Pharmacodynamic parameter

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No